CLINICAL TRIAL: NCT06991582
Title: Clinical Assessment of Injectable Composite Versus Packable Composite in Treatment of Carious Primary Anterior Teeth: A Randomized Clinical Trial
Brief Title: Clinical Assessment of Injectable Composite Versus Packable Composite in Treatment of Carious Primary Anterior Teeth
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Bassant Mohamed Elmesbahy, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 14422023595700
Record Dates: First submitted 2025-05-04; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Carious Primary; Carious Anteriors

STUDY DESIGN:
Intervention Model Description: Patients will be recruited from outpatient clinic of Pediatric Dentistry and Dental Public Health Department, Faculty of Dentistry Cairo University. Patients will be carefully assessed for eligibility to participate in our study then a full explanation of the nature of our experiment will be provided for parents or guardian before obtaining the informed consent from them.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Injectable composite (Experimental): Injectable composite Beautifil flow Plus X (Shofu INC., Koyoto, Japan)
  Interventions: Biological: Injectable composite resin restoration
- Packable Composite (Active Comparator): Packable Composite Beautifil II (Shofu INC., Koyoto, Japan)
  Interventions: Biological: packable composite

INTERVENTIONS:
Biological: Injectable composite resin restoration — Injectable composite Beautifil flow Plus X (Shofu INC., Koyoto, Japan)
  Arms: Injectable composite
Biological: packable composite — Packable Composite Beautifil II (Shofu INC., Koyoto, Japan)
  Arms: Packable Composite

SUMMARY:
The aim of this study is to evaluate the clinical success of injectable composite versus packable composite in restoration of primary anteriors.

ELIGIBILITY:
Inclusion Criteria:

* Children with caries in primary anterior teeth.
* Caries involving class III, IV, V or multisurface caries
* Restorable anterior teeth
* Pre operative Radiograph showing at least half of the root is not resorbed).

Exclusion Criteria:

* Badly decayed non restorable anterior teeth
* Signs and symptoms of root resorption (more than half the root is resorbed)
* Presence of bony resorption
* Presence of pathological root resorption
* Tooth Mobility

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2025-05-28 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Direct Clinical Assessment of Restoration | through study completion, on average of 1 year
  Modified United States Public Health Service (USPHS) Ryge Criteria Outcome name: Marginal integrity Measuring Device: Explorer
  Measuring unit:
  Alpha (A) There is no visible evidence of ditching along the margin of the restoration.
  Bravo (B) There is visible evidence of ditching along the margin of the restoration, it is not extending to the dentino-enamel junction.
  Charlie (C) There is dentin or base is exposed along the margin of the restoration.
  Delta (D) The restoration is mobile, fractured, or missing.
Direct Clinical Assessment of Restoration | through study completion, on average of 1 year
  Modified United States Public Health Service (USPHS) Ryge Criteria Outcome name: Color Match Measuring Device: Visual Inspection
  Measuring unit:
  Alpha (A) The restoration appears to match the shade and translucency of adjacent tooth tissues.
  Bravo (B)The restoration does not match the shade and translucency of adjacent tooth tissues, but the mismatch is within the normal range of tooth shades.
  Charlie (C)The restoration does not match the shade and translucency of the adjacent tooth structure, and the mismatch is outside the normal range of tooth shades and translucency
Direct Clinical Assessment of Restoration | through study completion, on average of 1 year
  Modified United States Public Health Service (USPHS) Ryge Criteria Outcome name: Cavo surface marginal discoloration Measuring Device: Visual Inspection
  Measuring unit:
  Alpha (A) There is no visual evidence of marginal discoloration different from the color of the restorative material and from the color of the adjacent tooth structure.
  Bravo (B) There is visual evidence of marginal discoloration at the junction of the tooth structure and the restoration, but the discoloration has not penetrated along the restoration in a pulpal direction.
  Charlie (C) There is visual evidence of marginal discoloration at the junction of the tooth structure and the restoration that has penetrated along the restoration in a pulpal direction.
Direct Clinical Assessment of Restoration | through study completion, on average of 1 year
  Modified United States Public Health Service (USPHS) Ryge Criteria Outcome name: Secondary Caries Measuring Device: Visual Inspection
  Measuring unit:
  Alpha (A) The restoration is a continuation of existing anatomic form adjacent to the restoration. Bravo (B) There is visual evidence of dark keep discoloration adjacent to the restoration (but not directly associated with cavosurface margins)
Direct Clinical Assessment of Restoration | through study completion, on average of 1 year
  Modified United States Public Health Service (USPHS) Ryge Criteria Outcome name: Anatomic Contour Measuring Device: Visual Inspection and Explorer
  Measuring unit:
  Alpha (A) Visual inspection and explorer The restoration is a continuation of existing anatomic form or is slightly flattened. It may be overcontoured. When the side of the explorer is placed tangentially across the restoration, it does not touch two opposing cavosurface line angles at the same time.
  Bravo (B) A surface concavity is evident. When the side of the explorer is placed tangentially across the restoration, it does not touch two opposing cavosurface line angles at the same time, but the dentin or base is not exposed.
  Charlie (C) There is a loss of restorative substance such that a surface concavity is evident and the base and/or dentin is exposed.
Direct Clinical Assessment of Restoration | through study completion, on average of 1 year
  Modified United States Public Health Service (USPHS) Ryge Criteria Outcome name: Surface Texture Measuring Device: Explorer
  Measuring unit:
  Alpha (A) Explorer Surface texture similar to polished enamel as determined by means of a sharp explorer.
  Bravo (B) Explorer Surface texture gritty or similar to a surface subjects to a white stone or similar to a composite containing supramicron-sized particles.
  Charlie (C) Explorer Surface pitting is sufficiently coarse to inhibit the continuous movement of an explorer across the surface.
Direct Clinical Assessment of Restoration | through study completion, on average of 1 year
  Modified United States Public Health Service (USPHS) Ryge Criteria Outcome name: Gross Fracture Measuring Device: Visual Inspection
  Measuring unit:
  Alpha (A) Restoration is intact and fully retained. Bravo (B) Restoration is partially retained with some portion of the restoration still intact.
  Charlie (C) Restoration is completely missing.

SECONDARY OUTCOMES:
Parents' patient Satisfaction | immediately after the intervention/procedure
  Measuring Device: Questionnaire Measuring unit: Binary (yes or No)
Chair side time | immediately after the intervention/procedure
  Measuring Device: Stopwatch Measuring unit: Minutes
Plaque accumulation | through study completion, on average of 1 year
  Measuring Device: Plaque index Score by Probe
  Measuring unit:
  0 : No plaque
  1. : A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may be seen in situ only by using the probe on the tooth surface.
  2. : Moderate accumulation of soft deposits within the gingival pocket, or the tooth and gingival margin which can be seen with the naked eye.
  3. : Abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin.

CONTACTS AND LOCATIONS:
Locations (1):
- Pediatric Dentistry Department, Faculty of Dentistry, Cairo University, Cairo, Egypt